CLINICAL TRIAL: NCT06037941
Title: Breathprinting (E-Nose) Technology to Measure Response to Treatment of Malignant Pleural Mesothelioma (MPM) Through MPM-Specific Volatile Organic Compounds Detected in Exhalates
Brief Title: Using E-Nose Technology to Measure Response to Treatment in People With Malignant Pleural Mesothelioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: UNIVERSITY CAMPUS BIO-MEDICO, ITALY (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-100
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Breathprinting (E-Nose) Technology; MPM-Specific Volatile Organic Compounds; 23-100
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-Nose Technology (Experimental): Patients undergo a breathprinting test (E-Nose) at baseline and at the first three standard of care follow-ups, as scheduled by their treating physician, that involve a CT of the Chest and/or PET/CT. The E-Nose testing will be administered by trained staff. Staff will use proper personal protective equipment during collections. Subjects will undergo E-Nose testing in a presurgical or interventional radiology suite. Subjects must consent to no smoking, no tooth brushing, and no food or drinks starting on midnight of the day of the E-Nose test. If fasting from midnight until the E-Nose test is not feasible, subjects may consent to fasting for 2 hours prior to each E-Nose test. Subjects opting to fast for 2 hours before each E-Nose test can only have still, non-carbonated water and non-aromatic foods or foods that do not develop aromatic compounds, such as low salt simple crackers, starting at midnight on the day of the E-Nose test until 2 hours before the collection.
  Interventions: Diagnostic Test: E-Nose testing; Diagnostic Test: Research blood

INTERVENTIONS:
Diagnostic Test: E-Nose testing — At baseline (before any treatment is administered) approximately when the patient is scheduled for a CT of the Chest and/or PET/CT after initiation of any treatment, as medically permissible and at the PI's discretion. A breath sample from each patient will be captured in a cartridge, which will form the basis for the E-Nose analysis, to be performed by study investigators at UCB.
Diagnostic Test: Research blood — Research blood tests will be obtained at baseline and the first three standard of care follow up visits, scheduled by their treating physician along with a CT of the Chest and/or PET/CT1 to determine whether serum biomarkers of MPM.

SUMMARY:
The researchers are doing this study to test the ability of a new technology called breathprinting, or electronic nose (E-Nose), to measure how people respond to standard treatment for malignant pleural mesothelioma (MPM). The researchers will study how E-Nose breathprints change over time as people receive standard treatment for MPM. They will also look at how changes in people's E-Nose breathprints compare to changes in their standard imaging scans and in biomarkers of MPM in their blood.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-85 years
* No history of thoracic cancer or extrathoracic cancer potentially involving pleural metastases (i.e., breast, gastric, colon, or pancreas cancer)
* Recent diagnosis of MPM
* Documented, signed, and dated informed consent, obtained before any procedures, for the proposed research study, and signed standard surgical consent for surgical resection

Exclusion Criteria:

* Aged <30 or >85 years at the first outpatient visit
* History of thoracic or extrathoracic cancer that puts the subject at risk for pleural or pulmonary metastases

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change of MPMspecific VOCs | up to 1 year
  compared with imaging (using RECIST 1.1 and mRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Rocco, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm